CLINICAL TRIAL: NCT02184624
Title: An Open-label Study of Inhaler Device Attributes Investigating Critical and Overall Errors, Ease of Use, and Preference Between a Number of Inhaler Devices (ELLIPTA, TURBUHALER, HANDIHALER, BREEZHALER, MDI, and DISKUS/ACCUHALER) in Adult Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study of Inhaler Device Attributes Investigating Critical and Overall Errors, Ease of Use, and Preference Between a Number of Inhaler Devices
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 200301
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: BREEZHALER; DISKUS/ACCUHALER; MDI; Inhaler preference; Overall inhaler error; HANDIHALER; Ease of use; TURBUHALER; ELLIPTA; Critical inhaler error
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Sub-Study 1 (Experimental): Subjects will be randomized to either use ELLIPTA inhaler first and then DISKUS/ACCUHALER inhaler or use DISKUS/ACCUHALER inhaler first and then ELLIPTA inhaler.
  Interventions: Device: ELLIPTA; Device: DISKUS/ACCUHALER
- Sub-Study 2 (Experimental): Subjects will be randomized to either use ELLIPTA inhaler first and then MDI inhaler or use MDI inhaler first and then ELLIPTA inhaler.
  Interventions: Device: ELLIPTA; Device: MDI
- Sub-Study 3 (Experimental): Subjects will be randomized to either use ELLIPTA inhaler first and then TURBUHALER inhaler or use TURBUHALER inhaler first and then ELLIPTA.
  Interventions: Device: ELLIPTA; Device: TURBUHALER
- Sub-Study 4 (Experimental): Subjects will be randomized to either use ELLIPTA inhaler first and then HANDIHALER inhaler or use HANDIHALER inhaler first and then ELLIPTA inhaler.
  Interventions: Device: ELLIPTA; Device: HANDIHALER
- Sub-Study 5 (Experimental): Subjects will be randomized to either use ELLIPTA inhaler first and then BREEZEHALER inhaler or use BREEZEHALER inhaler first and then ELLIPTA inhaler.
  Interventions: Device: ELLIPTA; Device: BREEZEHALER

INTERVENTIONS:
Device: ELLIPTA — Dry powder inhaler (placebo) with two blister strips. One placebo strip containing lactose monohydrate and a second placebo strip containing lactose monohydrate blended with magnesium stearate.
Device: DISKUS/ACCUHALER — Placebo inhaler with one blister strip containing lactose monohydrate.
  Arms: Sub-Study 1
Device: MDI — Placebo inhaler containing propellant (1,1,1, 2-Tetrafluoroethane).
  Arms: Sub-Study 2
Device: TURBUHALER — Placebo inhaler containing lactose monohydrate.
  Arms: Sub-Study 3
Device: HANDIHALER — Placebo inhaler containing lactose monohydrate in a capsule.
  Arms: Sub-Study 4
Device: BREEZEHALER — Placebo inhaler containing lactose monohydrate in a capsule.
  Arms: Sub-Study 5

SUMMARY:
This is a randomised, open-label, placebo, crossover, multicentre study with a single visit. The study will comprise five sub-studies. Subjects will receive inactive treatment (placebo) via the ELLIPTA® inhaler and one of the other inhaler devices depending on the sub-study they are randomised to. Only subjects who are naïve to the ELLIPTA inhaler and to one of the other inhaler devices that will be used in this study will be included. Furthermore, subjects who are naïve to the BREEZEHALER® and HANDIHALER® inhalers must be naïve to all other inhaler devices that requires a capsule. The study will be conducted in the UK and the Netherlands, and comprises one visit only. A sufficient number of subjects (at least 600) with COPD will be screened and 570 will be randomised to one of five sub-studies. Eligible subjects will be allocated to one of the sub-studies depending on their experience of using the other inhaler (i.e., depending on which other inhaler they are naïve to).

This study is designed to assess the proportion of COPD subjects making critical and overall (i.e., critical and non-critical errors) errors in using ELLIPTA inhaler and other commercially available inhaler devices such as the TURBUHALER®, HANDIHALER, BREEZHALER, MDI and DISKUS®/ACCUHALER® inhalers. This study will also assess the 'ease of use' and preference between the ELLIPTA inhaler and the other commercially available inhaler devices.

ELLIPTA, DISKUS, and ACCUHALER are registered trademarks of the GSK group of companies. TURBUHALER is a registered trademark of AstraZeneca. HANDIHALER is a registered trademark of Boehringer Ingelheim Pharma GmbH & Co. KG. BREEZHALER is a registered trademark of Novartis AG.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: Subject must give their signed and dated written informed consent to participate in the study; Subject understands and is willing, able, and likely to comply with study procedures and restrictions; Subject must be able to read, comprehend, and record information in Dutch and/or English.
* Age: >=40 years of age
* Gender: Male or female subjects.
* Primary diagnosis of COPD: subjects with a clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society. Comorbidities (rheumatoid arthritis or other locomotor problems, visual impairment, and depression or anxiety) will be documented as relevant to inhaler use.
* COPD treatment: All patients should be currently receiving treatment for COPD.
* Must be naïve to using ELLIPTA inhaler and at least one other inhaler device. Subjects who are naïve to the BREEZEHALER and HANDIHALER inhalers must be naïve to all other inhaler devices that requires a capsule.

Exclusion Criteria:

* Asthma: Subjects with a current diagnosis of asthma only. Note: Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD.
* Contraindications: A history of allergy or hypersensitivity to lactose/milk protein or magnesium stearate or to any other excipient.
* Subjects who are currently participating in another randomised pharmacological interventional trial.
* Inability to Read: In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a questionnaire and understand verbal instructions.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Netherlands (6):
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Beek
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Kloosterhaar
  - GSK Investigational Site, Nijverdal
  - GSK Investigational Site, Zutphen
- United Kingdom (2):
  - GSK Investigational Site, Portsmouth
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] van der Palen J, Thomas M, Chrystyn H, Sharma RK, van der Valk PD, Goosens M, Wilkinson T, Stonham C, Chauhan AJ, Imber V, Zhu CQ, Svedsater H, Barnes NC. A randomised open-label cross-over study of inhaler errors, preference and time to achieve correct inhaler use in patients with COPD or asthma: comparison of ELLIPTA with other inhaler devices. NPJ Prim Care Respir Med. 2016 Nov 24;26:16079. doi: 10.1038/npjpcrm.2016.79. PMID 27883002
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 200301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 28 August 2014 and 31 July 2015 at 8 centers, 6 in the Netherlands and 2 in the United Kingdom. Only participants who were naïve to the ELLIPTA inhaler and to one of the other inhaler devices that was used in this study were included.
Pre-assignment Details: A total of 575 participants were enrolled in the study out of them 8 failed in screening and remaining 567 were randomized and included in intent to treat population. Participants were allocated to a particular sub-study depending on their experience of using the other inhaler (i.e., depending on which other inhaler they were naïve to using).
Groups:
- Sub-study 1:ELLIPTA Versus (Vs) DISKUS/ACCUHALER: Participants received placebo via the ELLIPTA inhaler first and then DISKUS/ACCUHALER or DISKUS/ACCUHALER first and then ELLIPTA on Day 1. Participants continued to use their usual daily Chronic Obstructive Pulmonary Disease (COPD) maintenance and other medication(s) during the study.
- Sub-study 2: ELLIPTA Vs Metered-dose Inhaler (MDI): Participants received placebo via the ELLIPTA inhaler first and then MDI or MDI first and then ELLIPTA on Day 1. Participants continued to use their usual daily COPD maintenance and other medication(s) during the study.
- Sub-study 3: ELLIPTA Vs TURBUHALER: Participants received placebo via the ELLIPTA inhaler first and then TURBUHALER or TURBUHALER first and then ELLIPTA on Day 1. Participants continued to use their usual daily COPD maintenance and other medication(s) during the study.
- Sub-study 4: ELLIPTA Vs HANDIHALER: Participants received placebo via the ELLIPTA inhaler first and then HANDIHALER or HANDIHALER first and then ELLIPTA on Day 1. Participants continued to use their usual daily COPD maintenance and other medication(s) during the study.
- Sub-study 5: ELLIPTA Vs BREEZHALER: Participants received placebo via the ELLIPTA inhaler first and then BREEZHALER or BREEZHALER first and then ELLIPTA on Day 1. Participants continued to use their usual daily COPD maintenance and other medication(s) during the study.
Period: Overall Study
Arm/Group | Sub-study 1:ELLIPTA Versus (Vs) DISKUS/ACCUHALER | Sub-study 2: ELLIPTA Vs Metered-dose Inhaler (MDI) | Sub-study 3: ELLIPTA Vs TURBUHALER | Sub-study 4: ELLIPTA Vs HANDIHALER | Sub-study 5: ELLIPTA Vs BREEZHALER
Started | 171 | 80 | 100 | 118 | 98
Completed | 171 | 80 | 100 | 118 | 98
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER: Participants received placebo via the ELLIPTA inhaler first and then DISKUS/ACCUHALER or DISKUS/ACCUHALER first and then ELLIPTA on Day 1. Participants continued to use their usual daily COPD maintenance and other medication(s) during the study.
- Sub-study 2: ELLIPTA Vs MDI: Participants received placebo via the ELLIPTA inhaler first and then MDI or MDI first and then ELLIPTA on Day 1. Participants continued to use their usual daily COPD maintenance and other medication(s) during the study.
- Total: Total of all reporting groups
Arm/Group | Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER | Sub-study 2: ELLIPTA Vs MDI | Sub-study 3: ELLIPTA Vs TURBUHALER | Sub-study 4: ELLIPTA Vs HANDIHALER | Sub-study 5: ELLIPTA Vs BREEZHALER | Total
Number analyzed (Participants) | 171 | 80 | 100 | 118 | 98 | 567
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (7.41) | 65.6 (8.76) | 68.1 (8.66) | 67.3 (8.98) | 67.2 (8.17) | 67.3 (8.31)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 67 | 26 | 33 | 46 | 51 | 223
  Male | 103 | 53 | 67 | 72 | 47 | 342
  Unknown | 1 | 1 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 0 | 1 | 0 | 0 | 0 | 1
  Asian - East Asian Heritage | 0 | 1 | 0 | 0 | 0 | 1
  Asian - South East Asian Heritage | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 171 | 78 | 99 | 118 | 96 | 562
  Unknown | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Made at Least One Critical Error After Reading the Patient Information Leaflet
Description: A critical error was defined as an error that was most likely to result in no or only minimal medication being inhaled. The errors considered as critical errors while handling the inhaler devices were failed to open cover, lever was not pushed back, shook the device after dose preparation, exhaled directly into mouthpiece, no seal by the lips round the mouthpiece during the inhalation. As per the crossover study design participants received placebo via the ELLIPTA inhaler first and then non-ELLIPTA inhaler or non-ELLIPTA inhaler first and then ELLIPTA on Day 1. The percentage of participants who made at least one critical error was reported for each inhaler regardless sequence.
Time Frame: Day 1
Population: Modified Intent-to-Treat Population comprised of all participants in the Intent-to-Treat Population who completed demonstration of using both study inhaler devices after reading patient information leaflet.
Measure: Number; unit: Percentage of participants
Arm/Group | Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER | Sub-study 2: ELLIPTA Vs MDI | Sub-study 3: ELLIPTA Vs TURBUHALER | Sub-study 4: ELLIPTA Vs HANDIHALER | Sub-study 5: ELLIPTA Vs BREEZHALER
Number analyzed (Participants) | 171 | 80 | 100 | 118 | 98
Percentage of participants
  Error with only ELLIPTA inhaler | 2 | 4 | 1 | 4 | 8
  Error with only non-ELLIPTA inhaler | 40 | 51 | 37 | 38 | 41
  Error with both inhalers | 4 | 9 | 7 | 10 | 5
Statistical Analysis 1: Comparison: Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories Error while using only ELLIPTA inhaler Vs Error while using DISKUS/ACCUHALER
Statistical Analysis 2: Comparison: Sub-study 2: ELLIPTA Vs MDI; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using MDI
Statistical Analysis 3: Comparison: Sub-study 3: ELLIPTA Vs TURBUHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using TURBUHALER
Statistical Analysis 4: Comparison: Sub-study 4: ELLIPTA Vs HANDIHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using HANDIHALER
Statistical Analysis 5: Comparison: Sub-study 5: ELLIPTA Vs BREEZHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using BREEZHALER

2. Secondary Outcome: Percentage of Participants Who Made at Least One Overall Error After Reading the Patient Information Leaflet
Description: An overall error includes a critical and non-critical error. Any error made by the participants while demonstrating the use of the inhaler after reading the patient instruction leaflet was recorded by health care professional (HCP). The percentage of participants who made at least one overall error was reported. As per the crossover study design participants received placebo via the ELLIPTA inhaler first and then non-ELLIPTA inhaler or non-ELLIPTA inhaler first and then ELLIPTA on Day 1.
Time Frame: Day 1
Population: Modified Intent-to-Treat Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER | Sub-study 2: ELLIPTA Vs MDI | Sub-study 3: ELLIPTA Vs TURBUHALER | Sub-study 4: ELLIPTA Vs HANDIHALER | Sub-study 5: ELLIPTA Vs BREEZHALER
Number analyzed (Participants) | 171 | 80 | 100 | 118 | 98
Percentage of participants
  Error with only ELLIPTA inhaler | 10 | 1 | 5 | 10 | 8
  Error with only non-ELLIPTA inhaler | 45 | 55 | 45 | 29 | 34
  Error with both inhalers | 20 | 30 | 26 | 33 | 22
Statistical Analysis 1: Comparison: Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using DISKUS/ACCUHALER
Statistical Analysis 2: Comparison: Sub-study 2: ELLIPTA Vs MDI; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using MDI
Statistical Analysis 3: Comparison: Sub-study 3: ELLIPTA Vs TURBUHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using TURBUHALER
Statistical Analysis 4: Comparison: Sub-study 4: ELLIPTA Vs HANDIHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using HANDIHALER
Statistical Analysis 5: Comparison: Sub-study 5: ELLIPTA Vs BREEZHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using BREEZHALER

3. Secondary Outcome: Percentage of Participants Making at Least One Critical Error After the First Instruction From the HCP
Description: A critical error was defined as an error that was most likely to result in no or only minimal medication being inhaled. The errors considered as critical errors while handling the inhaler devices were failed to open cover, lever was not pushed back, shook the device after dose preparation, exhaled directly into mouthpiece, no seal by the lips round the mouthpiece during the inhalation. As per the crossover study design participants received placebo via the ELLIPTA inhaler first and then non-ELLIPTA inhaler or non-ELLIPTA inhaler first and then ELLIPTA on Day 1. If the participant made any error while demonstrating the use of the inhaler after reading the patient instruction leaflet, the HCP demonstrated the correct usage of the inhaler to the participant. The participants were then asked to demonstrate inhaler use again. If any further critical error were made by the participant, the error were recorded by HCP.
Time Frame: Day 1
Population: Modified Intent-to-Treat Population
Measure: Number; unit: Percentage of participants
Arm/Group | Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER | Sub-study 2: ELLIPTA Vs MDI | Sub-study 3: ELLIPTA Vs TURBUHALER | Sub-study 4: ELLIPTA Vs HANDIHALER | Sub-study 5: ELLIPTA Vs BREEZHALER
Number analyzed (Participants) | 171 | 80 | 100 | 118 | 98
Percentage of participants
  Error with only ELLIPTA inhaler | 0.6 | 4 | 0 | 0 | 1
  Error with only non-ELLIPTA inhaler | 2 | 15 | 10 | 17 | 11
  Error with both inhalers | 0.6 | 0 | 1 | 2 | 0
Statistical Analysis 1: Comparison: Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER; Test type: Superiority or Other; p = 0.480, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using DISKUS/ACCUHALER
Statistical Analysis 2: Comparison: Sub-study 2: ELLIPTA Vs MDI; Test type: Superiority or Other; p = 0.044, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using MDI
Statistical Analysis 3: Comparison: Sub-study 3: ELLIPTA Vs TURBUHALER; Test type: Superiority or Other; p = 0.025, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using TURBUHALER
Statistical Analysis 4: Comparison: Sub-study 4: ELLIPTA Vs HANDIHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using HANDIHALER
Statistical Analysis 5: Comparison: Sub-study 5: ELLIPTA Vs BREEZHALER; Test type: Superiority or Other; p = 0.014, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using BREEZHALER

4. Secondary Outcome: Percentage of Participants Making at Least One Overall Error After the First Instruction From the HCP
Description: An overall error includes a critical and non-critical error. If the participant made any error while demonstrating the use of the inhaler after reading the patient instruction leaflet, the HCP demonstrated the correct usage of the inhaler to the participant. The participants were then asked to demonstrate inhaler use again. If any further error was made by the participant was recorded by HCP.
Time Frame: Day 1
Population: Modified Intent-to-Treat Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER | Sub-study 2: ELLIPTA Vs MDI | Sub-study 3: ELLIPTA Vs TURBUHALER | Sub-study 4: ELLIPTA Vs HANDIHALER | Sub-study 5: ELLIPTA Vs BREEZHALER
Number analyzed (Participants) | 171 | 80 | 100 | 118 | 98
Percentage of participants
  Error with only ELLIPTA inhaler | 0.6 | 3 | 2 | 3 | 2
  Error with only non-ELLIPTA inhaler | 12 | 24 | 15 | 17 | 15
  Error with both inhalers | 4 | 1 | 4 | 8 | 0
Statistical Analysis 1: Comparison: Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using DISKUS/ACCUHALER
Statistical Analysis 2: Comparison: Sub-study 2: ELLIPTA Vs MDI; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using MDI
Statistical Analysis 3: Comparison: Sub-study 3: ELLIPTA Vs TURBUHALER; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using TURBUHALER
Statistical Analysis 4: Comparison: Sub-study 4: ELLIPTA Vs HANDIHALER; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using HANDIHALER
Statistical Analysis 5: Comparison: Sub-study 5: ELLIPTA Vs BREEZHALER; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — Statistical comparison for categories: Error while using only ELLIPTA inhaler Vs Error while using BREEZHALER

5. Secondary Outcome: Number of Participants Needed Instructions From HCP (Maximum Three Times) to Demonstrate Adequate Inhalation Technique
Description: If the participant made any error while demonstrating the use of the first inhaler after reading the patient instruction leaflet, the HCP demonstrated the correct usage of the inhaler to the participant. The participant was then asked to demonstrate inhaler use again. Any errors made by the participant were recorded by the HCP. The same procedure was repeated if the participant continues to make errors in the use of the inhaler. In total, the HCP demonstrated the use of the inhaler up to three times. Same procedure was followed for second inhaler. The number of participants who demonstrated the adequate inhalation technique after third time instructions from HCP was reported.
Time Frame: Day 1
Population: Modified Intent-to-Treat Population
Measure: Number; unit: Participants
Arm/Group | Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER | Sub-study 2: ELLIPTA Vs MDI | Sub-study 3: ELLIPTA Vs TURBUHALER | Sub-study 4: ELLIPTA Vs HANDIHALER | Sub-study 5: ELLIPTA Vs BREEZHALER
Number analyzed (Participants) | 171 | 80 | 100 | 118 | 98
Participants
  Zero HCP Instructions , ELLIPTA inhaler | 119 | 55 | 69 | 67 | 68
  Zero HCP Instructions , Non-ELLIPTA inhaler | 59 | 12 | 29 | 45 | 43
  One HCP Instructions , ELLIPTA inhaler | 45 | 22 | 25 | 38 | 28
  One HCP Instructions , Non-ELLIPTA inhaler | 85 | 48 | 52 | 44 | 40
  Two HCP Instructions , ELLIPTA inhaler | 5 | 2 | 4 | 8 | 0
  Two HCP Instructions , Non-ELLIPTA inhaler | 19 | 12 | 11 | 13 | 8
  Three HCP Instructions , ELLIPTA inhaler | 1 | 0 | 1 | 3 | 2
  Three HCP Instructions , Non-ELLIPTA inhaler | 4 | 2 | 1 | 6 | 4
Statistical Analysis 1: Comparison: Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test — Number of participants requiring instructions from the HCP (maximum three times) to demonstrate adequate inhalation technique of ELLIPTA inhaler versus those for DISKUS/ACCUHALER inhaler
Statistical Analysis 2: Comparison: Sub-study 2: ELLIPTA Vs MDI; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test — Number of participants requiring instructions from the HCP (maximum three times) to demonstrate adequate inhalation technique of ELLIPTA inhaler versus those for MDI inhaler
Statistical Analysis 3: Comparison: Sub-study 3: ELLIPTA Vs TURBUHALER; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test — Number of participants requiring instructions from the HCP (maximum three times) to demonstrate adequate inhalation technique of ELLIPTA inhaler versus those for TURBUHALER inhaler
Statistical Analysis 4: Comparison: Sub-study 4: ELLIPTA Vs HANDIHALER; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test — Number of participants requiring instructions from the HCP (maximum three times) to demonstrate adequate inhalation technique of ELLIPTA inhaler versus those for HANDIHALER inhaler
Statistical Analysis 5: Comparison: Sub-study 5: ELLIPTA Vs BREEZHALER; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test — Number of participants requiring instructions from the HCP (maximum three times) to demonstrate adequate inhalation technique of ELLIPTA inhaler versus those for BREEZHALER inhaler

6. Secondary Outcome: Percentage of Participants Who Overall Preferred the ELLIPTA Device Compared to Non-ELLIPTA Inhalers as Assessed by the Preference Questionnaire
Description: After completing the demonstration procedures of the inhalers, the HCP asked the participant a number of questions from preference questionnaire. Preference questionnaire consisted of eight questions related to both inhalers used during the study. Each question had one response to choose from 3 preference options (Other inhaler device, ELLIPTA inhaler device and No preference). The number of participants who overall preferred the ELLIPTA device compared to non-ELLIPTA inhalers (First question in the preference questionnaire) were reported.
Time Frame: Day 1
Population: Modified Intent-to-Treat population. Only participants who completed the questionnaire were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER | Sub-study 2: ELLIPTA Vs MDI | Sub-study 3: ELLIPTA Vs TURBUHALER | Sub-study 4: ELLIPTA Vs HANDIHALER | Sub-study 5: ELLIPTA Vs BREEZHALER
Number analyzed (Participants) | 170 | 80 | 100 | 118 | 98
Percentage of participants
  ELLIPTA preferred | 74 | 75 | 86 | 87 | 72
  Non-ELLIPTA Device Preferred | 11 | 19 | 6 | 11 | 19
  No preference | 15 | 6 | 8 | 2 | 8
Statistical Analysis 1: Comparison: Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Number of participants preferring ELLIPTA device versus number of participants preferring DISKUS/ACCUHALER device as assessed by the 'preference' questionnaire
Statistical Analysis 2: Comparison: Sub-study 2: ELLIPTA Vs MDI; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Number of participants preferring ELLIPTA device versus number of participants preferring MDI device as assessed by the 'preference' questionnaire
Statistical Analysis 3: Comparison: Sub-study 3: ELLIPTA Vs TURBUHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Number of participants preferring ELLIPTA device versus number of participants preferring TURBUHALER device as assessed by the 'preference' questionnaire
Statistical Analysis 4: Comparison: Sub-study 4: ELLIPTA Vs HANDIHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Number of participants preferring ELLIPTA device versus number of participants preferring HANDIHALER device as assessed by the 'preference' questionnaire
Statistical Analysis 5: Comparison: Sub-study 5: ELLIPTA Vs BREEZHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Number of participants preferring ELLIPTA device versus number of participants preferring BREEZHALER device as assessed by the 'preference' questionnaire

7. Secondary Outcome: Percentage of Participants Who Overall Found the ELLIPTA Device Easy to Use Compared With Non-ELLIPTA Inhalers as Assessed by the Ease of Use Questionnaire
Description: After completing the demonstration procedures of the inhalers, the HCP asked the participant a number of questions from ease of use questionnaire. Ease of use questionnaire consisted of six questions each for ELLIPTA inhaler and the other inhaler under study. Each question had one response to choose from 5 options of ease of use (Very easy, easy, neutral, difficult and very difficult). Based upon the response given by the participants the number of participants who rated ease of use higher for ELLIPTA, higher for non- ELLIPTA, or rated the same were reported
Time Frame: Day 1
Population: Modified Intent-to-Treat Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER | Sub-study 2: ELLIPTA Vs MDI | Sub-study 3: ELLIPTA Vs TURBUHALER | Sub-study 4: ELLIPTA Vs HANDIHALER | Sub-study 5: ELLIPTA Vs BREEZHALER
Number analyzed (Participants) | 171 | 80 | 100 | 118 | 98
Percentage of participants
  RATED HIGHER FOR ELLIPTA | 66 | 66 | 72 | 78 | 65
  RATED HIGHER FOR NON-ELLIPTA DEVICES | 5 | 10 | 4 | 2 | 12
  RATED SAME FOR BOTH TYPES | 29 | 24 | 24 | 20 | 22
Statistical Analysis 1: Comparison: Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Number of participants preferring ELLIPTA device versus number of participants preferring DISKUS/ACCUHALER device by the 'ease of use' questionnaire
Statistical Analysis 2: Comparison: Sub-study 2: ELLIPTA Vs MDI; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Number of participants preferring ELLIPTA device versus number of participants preferring MDI device by the 'ease of use' questionnaire
Statistical Analysis 3: Comparison: Sub-study 3: ELLIPTA Vs TURBUHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Number of participants preferring ELLIPTA device versus number of participants preferring TURBUHALER device by the 'ease of use' questionnaire
Statistical Analysis 4: Comparison: Sub-study 4: ELLIPTA Vs HANDIHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Number of participants preferring ELLIPTA device versus number of participants preferring HANDIHALER device by the 'ease of use' questionnaire
Statistical Analysis 5: Comparison: Sub-study 5: ELLIPTA Vs BREEZHALER; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Number of participants preferring ELLIPTA device versus number of participants preferring BREEZHALER device by the 'ease of use' questionnaire

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected from the start of study treatment (Day 1) and until the follow up contact.
Description: Intent-to-Treat Population comprised of all participants who had been randomized and used at least one study inhaler after reading patient information leaflet.
Arm/Group | Sub-study 1:ELLIPTA Vs DISKUS/ACCUHALER | Sub-study 2: ELLIPTA Vs MDI | Sub-study 3: ELLIPTA Vs TURBUHALER | Sub-study 4: ELLIPTA Vs HANDIHALER | Sub-study 5: ELLIPTA Vs BREEZHALER
Serious Adverse Events (participants affected / at risk) | 0/171 | 0/80 | 0/100 | 0/118 | 0/98
Other Adverse Events (participants affected / at risk) | 0/171 | 0/80 | 0/100 | 0/118 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.